CLINICAL TRIAL: NCT02394041
Title: A Randomised Controlled Multicenter Trial Evaluating the Efficacy of Acupuncture Versus Placebo on the Caesarean Section Rate in Case of Cervical Dystocia in Full-term Pregnancy
Brief Title: Randomised Controlled Trial of the Efficacy of Acupuncture Versus Placebo on the Caesarean Section Rate in Case of Cervical Dystocia in Full-term Pregnancy
Acronym: ACUCESAR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient recruitment: 142 patients instead of 2,220 planned
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P081233; AOM09091 (Other Grant/Funding Number: APHP)
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-02

CONDITIONS: Cervical Dystocia
Keywords: acupuncture; cervical dystocia; caesarean section; obstetric labor; randomized controlled trial
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- acupuncture (Experimental): The first session of acupuncture treatment will be performed at the inclusion visit, 2 additional acupuncture sessions will be scheduled as 1 session per week for the next 2 weeks.
  One or more additional session will be performed in the delivery room.
  Interventions: Device: Acupuncture
- Sham acupuncture (Sham Comparator): The same as active arm but with sham needles.
  Interventions: Device: Sham acupuncture
- control group (No Intervention): Standard care, no acupuncture session.

INTERVENTIONS:
Device: Acupuncture — Method of acupuncture: check the condition of skin, disinfect if needed, insert sterile needles with special handling for each point, remove the needles after 15 minutes.
  Arms: acupuncture
Device: Sham acupuncture — Sham acupuncture with sham needles
  Arms: Sham acupuncture

SUMMARY:
The principal objective of the trial is to demonstrate that acupuncture could reduce the caesarean section rate for cervical dystocia.

Secondary objectives:

To demonstrate that acupuncture can:

* reduce morbidity, fetal mortality and duration of childbirth;
* reduce the cost of care, due to diminution of caesarean sections and duration of obstetric labor;
* to evaluate the tolerance.

DETAILED DESCRIPTION:
In this trial, pregnant women with at least 37 weeks of amenorrhea will be randomized to traditional chinese acupuncture, sham acupuncture, or usual care only.

9 investigator sites will participate to this trial targeting to enrol 2220 patients in total. 1780 subjects will receive acupuncture treatment, either effective treatment or sham, whereas 400 patients will receive usual care only.

Acupuncture therapy consists in stimulations on specific skin points of the abdominal area, which are specific acupuncture points in traditional chinese medicine for the induction of obstetric labor, according to the professional recommendations of the French Acupuncture and Traditional Chinese Medicine College.

Each patient will have a 5-week follow-up in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Signed informed consent
* Woman carrying one foetus only
* at 37 weeks (+/- 2 days) of amenorrhea
* Without contraindication to vaginal delivery

Exclusion Criteria:

* Prior history of caesarean section
* Non-cephalic presentation
* Fetal macrosomia
* Multiple pregnancy
* Chronic fetal hypoxia
* Placenta praevia
* Risk of neonatal contamination

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2012-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Caesarean section rate | up to 37 weeks
  Rate of caesarean section for cervical dystocia in full-time pregnancies

CONTACTS AND LOCATIONS:
Overall Officials: Denis COLIN, MD, Principal Investigator — Department of Obstetrics, Hôpital Saint-Cloud
Locations (1):
- Department of Obstetrics, Hôpital Saint-Cloud, Saint-Cloud, Hauts-de-Seine, France